CLINICAL TRIAL: NCT07091864
Title: Phase II Randomized Trial Of Glucose Monitoring In Glioblastoma
Brief Title: Continuous Glucose Monitoring for the Management of Hyperglycemia in Patients With Glioblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SING; NCI-2025-04735 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-006112 (Other: Mayo Clinic Institutional Review Board); SING (Other: Mayo Clinic)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma, IDH-Wildtype; WHO Grade 4 Glioma
MeSH Terms: conditions — Glioblastoma | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Diet Therapy; Glucose; Magnetic Resonance Spectroscopy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To reduce bias, all imaging and quality of life assessments will be interpreted by evaluators blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (SOC, CGM) (Experimental): Patients receive SOC treatment plus CGM with endocrinology-guided interventions as needed and attend dietary counseling sessions once a month for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI throughout the trial.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Dietary Intervention; Procedure: Magnetic Resonance Imaging; Other: Monitoring; Other: Questionnaire Administration; Other: Supportive Care
- Arm B (SOC, intermittent glucose monitoring) (Active Comparator): Patients receive SOC treatment plus intermittent glucose monitoring as clinically indicated for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI throughout the trial.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Glucose Measurement; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC treatment
  Other Names: standard of care; standard therapy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Dietary Intervention — Attend dietary counseling sessions
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm A (SOC, CGM)
Other: Glucose Measurement — Undergo intermittent glucose monitoring
  Other Names: GLUC; Glucose
  Arms: Arm B (SOC, intermittent glucose monitoring)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Monitoring — Undergo CGM
  Other Names: monitor
  Arms: Arm A (SOC, CGM)
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive endocrinology-guided interventions
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Arm A (SOC, CGM)

SUMMARY:
This clinical trial studies whether continuous glucose monitoring (CGM) can be used to help patients with glioblastoma manage their blood sugar (glucose) levels and improve survival. Glioblastoma is the most common malignant primary brain tumor in adults, with an average survival time of approximately 15-18 months despite therapy. Studies have shown that having a higher-than-normal amount of glucose in the blood (hyperglycemia) during radiation therapy is associated with poorer survival outcomes in glioblastoma patients. Hyperglycemia in glioblastoma patients is often driven by steroids that are commonly used during treatment. CGM uses a device that places a sensor under the skin that monitors glucose levels at regular intervals, providing real-time, or near real-time, glucose information. This can help to identify when a patient has changes in their glucose levels so they may receive necessary interventions or medications sooner. CGM may be an effective way for glioblastoma patients to manage their glucose levels, which may improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Presumed newly diagnosed GBM based on imaging findings consistent with GBM on brain MRI (e.g., heterogeneously enhancing mass with central necrosis and surrounding edema), as determined by the treating neuro-oncology team
* Age ≥ 18 years at the time of consent
* Karnofsky performance status (KPS) ≥ 70 at baseline
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
* Platelet count ≥ 100 × 10^9/L
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN
* Total bilirubin ≤ 1.5 × ULN
* Willingness and ability to comply with CGM device use and attend dietary counseling sessions as part of the study protocol

Exclusion Criteria:

* Recurrent glioblastoma or prior therapy for glioblastoma beyond surgical resection or biopsy
* History of eating disorders (e.g., anorexia nervosa, bulimia) or substance use disorder within the past 12 months
* Any other uncontrolled or inadequately managed medical illness (e.g., unstable cardiovascular, hepatic, renal, or psychiatric condition) that, in the opinion of the investigator, would interfere with study participation or interpretation of results
* Concurrent diagnosis of another active malignancy requiring treatment
* Pregnancy or breastfeeding at the time of enrollment
* Documented history of type 1 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 12 months | At 12 months
  Defined as the time from study enrollment until death due to any cause.

SECONDARY OUTCOMES:
Incidence of symptomatic hypoglycemia | Up to 52 weeks
  Will be defined as continuous glucose monitoring glucose < 70 mg/dL with concurrent symptoms. Proportion of participants with ≥ 1 symptomatic hypoglycemia event will be analyzed with Fisher's exact test.
Quality of Life - EORTC QLQ C-30 | At baseline, 3 months, 6 months, and 12 months
  The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 is a 30-item questionnaire where 28 questions are answered on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, and 4= very much) and 2 two questions are answered on a scale of 1-7 (1= very poor and 7=excellent). Higher summary scores indicate better health related quality of life.
Quality of Life - EORTC QLQ-BN20 | At baseline, 3 months, 6 months, and 12 months
  The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-BN20 is a 20-item questionnaire related to symptoms experienced by patients with brain cancer during the past week. Questions are answered on a scale of 1-4 where 1=not at all, 2=a little; 3-quite a bit; and 4=very much. Higher scores indicate greater severity of symptoms.
Hemoglobin (HbA1c) | At 3 months, 6 months, and 12 months
  Compared at 3, 6 and 12 months using repeated measures mixed models. Model based contrasts will be used to estimate the between group changes from baseline in A1c values. Random intercept will be used.
Fasting glucose | At 3 months, 6 months, and 12 months
  Compared at 3, 6 and 12 months using repeated measures mixed models. Random intercept will be used.
Lactate levels (continuous) | At 3 months, 6 months, and 12 months
  Compared at 3, 6 and 12 months using repeated measures mixed models. Random intercept will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Zadeh, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials